CLINICAL TRIAL: NCT03914495
Title: The Role of Microbiome Reprogramming on Liver Fat Accumulation
Acronym: MILE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI carefully considered multiple factors and decided to close study to any further enrollment.
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1312439
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: NAFLD
Keywords: inulin; microbiome; hepatic steatosis; obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Obesity | interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive powdered maltodextrin to provide equivalent calories and macronutrients without any fiber.
  Interventions: Dietary Supplement: Placebo
- Inulin (Active Comparator): Participants will receive inulin, 10 grams TID for 28 days with titration as follows: 10 grams QD for 3 days, 20 grams BID for 4 days with the remaining 21 days at 10 g TID.
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Inulin — Powdered inulin will be provided in pre-weighed portions for consumption in a 1 week titration to reduce GI side effects with a 21 day intervention at full dose.
  Arms: Inulin
Dietary Supplement: Placebo — Powdered maltodextrin will be provided in pre-weighed portions for consumption in a 1 week titration with a 21 day intervention at full dose.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether reprogramming the microbiome via soluble fiber supplementation will decrease liver fat in obese individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35-65 years
2. Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF) 5%-30% (+0.5%)
3. Liver stiffness <3.5 kPa by Magnetic Resonance Elastography (MRE)
4. Body mass index (BMI) 27.5-45 kg/m2
5. Weight stable (weight change of no more than 3 kg +0.5 kg) during the 6 months prior to enrollment
6. For individuals with type 2 diabetes: HbA1c ≥6.5 - <9.5%. If taking allowable diabetes medications, HbA1c can be below 6.5%.
7. Fasting triglycerides 400 mg/dL (4.5 mmol/L)
8. Able to speak and understand written and spoken English
9. Understands the procedures and agrees to participate by giving written informed consent
10. Willing and able to comply with scheduled study days, laboratory tests, and other study procedures

Exclusion Criteria:

Acute or chronic medical conditions or medication that would contraindicate the participation in the research testing or could potentially affect metabolic function including, but not limited to:

1. Diagnosis of type 1 diabetes mellitus
2. Insulin use
3. Change within 3 months of screening of any medication used to treat insulin resistance or type 2 diabetes
4. History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males within the previous 6 months (1 drink = 5 ounces [150 mL] of wine, 12 ounces [360 mL] of beer, or 1.5 ounces [45 mL] of hard liquor)
5. A total score of 8 on the Alcohol Use Disorders Identification Test (AUDIT) questionnaire, indicating harmful or hazardous alcohol consumption
6. Clinical evidence of hepatic decompensation, including, but not limited to esophageal varices, ascites, or hepatic encephalopathy
7. Evidence of other forms of chronic liver disease (including laboratory tests and confirmed with a single repeat, if needed):

   * Hepatitis B virus: defined by presence of hepatitis B surface antigen
   * Hepatitis C virus: As defined by a clinical history of previous diagnosis of Hepatitis C (treated or untreated) or a positive Hepatitis C antibody.
   * Known diagnosis of primary biliary cirrhosis, primary sclerosing cholangitis, autoimmune hepatitis, or overlap syndrome
   * Alcoholic liver disease
   * Known diagnosis of hemochromatosis
   * Prior known drug-induced liver injury
   * Known or suspected hepatocellular carcinoma or other liver cancer
   * History of liver transplant, current placement on a liver transplant list, or current model of end-stage liver disease (MELD) score >12
   * Histological presence of cirrhosis on a prior biopsy
8. Bleeding disorders
9. Acute or chronic infections
10. Severe asthma or chronic obstructive pulmonary disease
11. Renal insufficiency or nephritis
12. Thyroid dysfunction (suppressed TSH, elevated TSH <10 µIU/ml if symptomatic or elevated TSH >10 µIU/ml if asymptomatic)
13. Uncontrolled hypertension (BP >160 mmHg systolic or >100 mmHg diastolic)
14. Prior or planned bariatric surgery
15. Gastrointestinal disorders including: inflammatory bowel disease or malabsorption, swallowing disorders, suspected or known strictures, fistulas or physiological/mechanical GI obstruction, history of gastrointestinal surgery, Crohn's disease or diverticulitis.
16. Participants with intolerance to soluble fiber, sucralose or erythritol.
17. A positive urine drug test for illicit drugs
18. History of major depression within <5 years from screening or which, in the opinion of a medical investigator, will impact the participant's ability to complete the study.
19. History of eating disorders
20. History of Cushing's disease or syndrome
21. Untreated or inadequately controlled hypo- or hyperthyroidism
22. Active rheumatoid arthritis or other inflammatory rheumatic disorder
23. Pregnant or nursing females or females less than 6 months postpartum from the scheduled date of collection
24. Nicotine use within the past 3 months
25. Had major surgery within 4 weeks prior to Screening.
26. Anemia (hemoglobin <12 g/dl in men, <11 g/dl in women) during screening
27. Participation in studies involving investigational drug(s) within 30 days prior to Screening
28. History or presence of cardiovascular disease (unstable angina, myocardial infarction or coronary revascularization within 6 months, presence of cardiac pacemaker, implanted cardiac defibrillator)
29. Human Immunodeficiency Virus (HIV) infection defined as: previous diagnosis of HIV infection, history of positive screening or quantitative HIV testing; positive HIV screen
30. Any malignancy not considered cured, except basal cell carcinoma and squamous cell carcinoma of the skin (a participant is considered cured if there has been no evidence of cancer recurrence in the previous 5 years)
31. Use of drugs historically associated with non-alcoholic fatty liver disease (NAFLD) for 1 month in the previous year prior to Screening; examples include: amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, other known hepatotoxins
32. Participants who fulfill any of the contraindications for MRI; examples include metal implants, devices, paramagnetic objects contained within the body and excessive or metal-containing tattoos
33. Unable to participate in MR assessments due to physical limitations or equipment tolerances (e.g., MRI bore size and 500-pound weight limit) based on Investigator's judgment at screening
34. Any person with history of severe claustrophobia or unable to lie still within the environment of the MRI scanner or unable maintain a breath hold for the required period to acquire images without mild sedation/treatment with an anxiolytic
35. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to Screening (participants may not donate blood any time during the study, through the final study day)
36. Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete study days

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Absolute Change in Liver Fat | 28 days
  Liver fat changes will be assessed by MRI-PDFF

CONTACTS AND LOCATIONS:
Overall Officials: Karen Corbin, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

REFERENCES:
- [Background] Estes C, Razavi H, Loomba R, Younossi Z, Sanyal AJ. Modeling the epidemic of nonalcoholic fatty liver disease demonstrates an exponential increase in burden of disease. Hepatology. 2018 Jan;67(1):123-133. doi: 10.1002/hep.29466. Epub 2017 Dec 1. PMID 28802062
- [Background] Rinella ME. Nonalcoholic fatty liver disease: a systematic review. JAMA. 2015 Jun 9;313(22):2263-73. doi: 10.1001/jama.2015.5370. PMID 26057287
- [Background] Cohen JC, Horton JD, Hobbs HH. Human fatty liver disease: old questions and new insights. Science. 2011 Jun 24;332(6037):1519-23. doi: 10.1126/science.1204265. PMID 21700865
- [Background] Stefan N, Haring HU, Cusi K. Non-alcoholic fatty liver disease: causes, diagnosis, cardiometabolic consequences, and treatment strategies. Lancet Diabetes Endocrinol. 2019 Apr;7(4):313-324. doi: 10.1016/S2213-8587(18)30154-2. Epub 2018 Aug 30. PMID 30174213
- [Background] Caputo T, Gilardi F, Desvergne B. From chronic overnutrition to metaflammation and insulin resistance: adipose tissue and liver contributions. FEBS Lett. 2017 Oct;591(19):3061-3088. doi: 10.1002/1873-3468.12742. Epub 2017 Jul 25. PMID 28677122
- [Background] Younossi Z, Anstee QM, Marietti M, Hardy T, Henry L, Eslam M, George J, Bugianesi E. Global burden of NAFLD and NASH: trends, predictions, risk factors and prevention. Nat Rev Gastroenterol Hepatol. 2018 Jan;15(1):11-20. doi: 10.1038/nrgastro.2017.109. Epub 2017 Sep 20. PMID 28930295
- [Background] Valbusa F, Agnoletti D, Scala L, Grillo C, Arduini P, Bonapace S, Calabria S, Scaturro G, Mantovani A, Zoppini G, Turcato E, Maggioni AP, Arcaro G, Targher G. Non-alcoholic fatty liver disease and increased risk of all-cause mortality in elderly patients admitted for acute heart failure. Int J Cardiol. 2018 Aug 15;265:162-168. doi: 10.1016/j.ijcard.2018.04.129. Epub 2018 May 2. PMID 29739707
- [Background] Adams LA, Harmsen S, St Sauver JL, Charatcharoenwitthaya P, Enders FB, Therneau T, Angulo P. Nonalcoholic fatty liver disease increases risk of death among patients with diabetes: a community-based cohort study. Am J Gastroenterol. 2010 Jul;105(7):1567-73. doi: 10.1038/ajg.2010.18. Epub 2010 Feb 9. PMID 20145609
- [Background] Fabbrini E, Magkos F, Mohammed BS, Pietka T, Abumrad NA, Patterson BW, Okunade A, Klein S. Intrahepatic fat, not visceral fat, is linked with metabolic complications of obesity. Proc Natl Acad Sci U S A. 2009 Sep 8;106(36):15430-5. doi: 10.1073/pnas.0904944106. Epub 2009 Aug 24. PMID 19706383
- [Background] Lonardo A, Sookoian S, Pirola CJ, Targher G. Non-alcoholic fatty liver disease and risk of cardiovascular disease. Metabolism. 2016 Aug;65(8):1136-50. doi: 10.1016/j.metabol.2015.09.017. Epub 2015 Sep 25. PMID 26477269
- [Background] Loomba R, Sanyal AJ, Kowdley KV, Terrault N, Chalasani NP, Abdelmalek MF, McCullough AJ, Shringarpure R, Ferguson B, Lee L, Chen J, Liberman A, Shapiro D, Neuschwander-Tetri BA. Factors Associated With Histologic Response in Adult Patients With Nonalcoholic Steatohepatitis. Gastroenterology. 2019 Jan;156(1):88-95.e5. doi: 10.1053/j.gastro.2018.09.021. Epub 2018 Sep 15. PMID 30222962
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] Dumas ME, Barton RH, Toye A, Cloarec O, Blancher C, Rothwell A, Fearnside J, Tatoud R, Blanc V, Lindon JC, Mitchell SC, Holmes E, McCarthy MI, Scott J, Gauguier D, Nicholson JK. Metabolic profiling reveals a contribution of gut microbiota to fatty liver phenotype in insulin-resistant mice. Proc Natl Acad Sci U S A. 2006 Aug 15;103(33):12511-6. doi: 10.1073/pnas.0601056103. Epub 2006 Aug 8. PMID 16895997
- [Background] Zhou D, Pan Q, Shen F, Cao HX, Ding WJ, Chen YW, Fan JG. Total fecal microbiota transplantation alleviates high-fat diet-induced steatohepatitis in mice via beneficial regulation of gut microbiota. Sci Rep. 2017 May 8;7(1):1529. doi: 10.1038/s41598-017-01751-y. PMID 28484247
- [Background] Le Roy T, Llopis M, Lepage P, Bruneau A, Rabot S, Bevilacqua C, Martin P, Philippe C, Walker F, Bado A, Perlemuter G, Cassard-Doulcier AM, Gerard P. Intestinal microbiota determines development of non-alcoholic fatty liver disease in mice. Gut. 2013 Dec;62(12):1787-94. doi: 10.1136/gutjnl-2012-303816. Epub 2012 Nov 29. PMID 23197411
- [Background] Kaden-Volynets V, Basic M, Neumann U, Pretz D, Rings A, Bleich A, Bischoff SC. Lack of liver steatosis in germ-free mice following hypercaloric diets. Eur J Nutr. 2019 Aug;58(5):1933-1945. doi: 10.1007/s00394-018-1748-4. Epub 2018 Jun 20. PMID 29926176
- [Background] De Minicis S, Rychlicki C, Agostinelli L, Saccomanno S, Candelaresi C, Trozzi L, Mingarelli E, Facinelli B, Magi G, Palmieri C, Marzioni M, Benedetti A, Svegliati-Baroni G. Dysbiosis contributes to fibrogenesis in the course of chronic liver injury in mice. Hepatology. 2014 May;59(5):1738-49. doi: 10.1002/hep.26695. Epub 2014 Feb 25. PMID 23959503
- [Background] Kang DJ, Betrapally NS, Ghosh SA, Sartor RB, Hylemon PB, Gillevet PM, Sanyal AJ, Heuman DM, Carl D, Zhou H, Liu R, Wang X, Yang J, Jiao C, Herzog J, Lippman HR, Sikaroodi M, Brown RR, Bajaj JS. Gut microbiota drive the development of neuroinflammatory response in cirrhosis in mice. Hepatology. 2016 Oct;64(4):1232-48. doi: 10.1002/hep.28696. Epub 2016 Jul 29. PMID 27339732
- [Background] Mazagova M, Wang L, Anfora AT, Wissmueller M, Lesley SA, Miyamoto Y, Eckmann L, Dhungana S, Pathmasiri W, Sumner S, Westwater C, Brenner DA, Schnabl B. Commensal microbiota is hepatoprotective and prevents liver fibrosis in mice. FASEB J. 2015 Mar;29(3):1043-55. doi: 10.1096/fj.14-259515. Epub 2014 Dec 2. PMID 25466902
- [Background] Henao-Mejia J, Elinav E, Jin C, Hao L, Mehal WZ, Strowig T, Thaiss CA, Kau AL, Eisenbarth SC, Jurczak MJ, Camporez JP, Shulman GI, Gordon JI, Hoffman HM, Flavell RA. Inflammasome-mediated dysbiosis regulates progression of NAFLD and obesity. Nature. 2012 Feb 1;482(7384):179-85. doi: 10.1038/nature10809. PMID 22297845
- See also: Webpage for Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org